CLINICAL TRIAL: NCT04946032
Title: Optimum Length of Catheter in the Epidural Space for Labor Analgesia in Non-obese Women: a Randomised Controlled Trial of 4 Cm Versus 5 Cm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-06
Record Dates: First submitted 2021-06-25; First posted 2021-06-30 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Labor Pain
Keywords: epidural catheter; epidural analgesia; labor epidural
MeSH Terms: conditions — Labor Pain | interventions — Injections, Epidural

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist placing the epidural will know the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 cm epidural catheter (Active Comparator): The epidural catheter will be thread into the epidural space at a length of 4 cm.
  Interventions: Other: Epidural catheter
- 5 cm epidural catheter (Active Comparator): The epidural catheter will be thread into the epidural space at a length of 5 cm.
  Interventions: Other: Epidural catheter

INTERVENTIONS:
Other: Epidural catheter — The epidural catheter length will vary, either 4 cm or 5 cm into the epidural space.
  Other Names: epidural

SUMMARY:
Epidural analgesia was introduced to the world of obstetrics in 1909 by Walter Stoeckel. Over the following 100 years it has developed to become the gold-standard for delivery of intra-partum analgesia, with between 60 and 75% of North American parturients receiving an epidural during their labor. Effective labor analgesia has been shown to improve maternal and fetal outcomes. One aspect of catheter insertion that has not been fully evaluated, and with very little recent work undertaken, is the optimal length of epidural catheter to be left in the epidural space. Dislodgement or displacement of epidural catheter remains a significant cause for failure with analgesia. Novel methods of fixation may further reduce the risk of catheter migration. Another factor is the direction of travel within the epidural space, only 13% of lumbar catheters remain uncoiled after insertion of more than 4 cm into the epidural space.

Hypothesis: The investigators hypothesize that catheters inserted to 4 cm will have a lower rate of failure when compared to those inserted to 5 cm.

Objective: This study aims to evaluate the difference in quality of labor analgesia delivered by epidural catheters inserted to either 4 or 5 cm into the epidural space.

This study will be conducted as an interventional double-blinded randomised control trial to establish best practice.

DETAILED DESCRIPTION:
Effective labor analgesia has been shown to improve maternal and fetal outcomes. It is of paramount importance to the obstetric anesthesiologist to optimize the quality of labor analgesia and identify any factors leading to ineffective epidural analgesia. One aspect of catheter insertion that has not been fully evaluated, and with very little recent work undertaken, is the optimal length of epidural catheter to be left in the epidural space.

Previous studies have advocated, for varying reasons, different lengths of catheter to be left in the space; these range from 2cm to 8cm. Longer epidural lengths in the space can be associated with foraminal escape, leading to unilateral block, and intravascular insertion, prompting additional manipulation. Shorter lengths have previously been associated with more frequent dislodgement. The directionality of the epidural catheter once in the space has been demonstrated to correlate with misdirection.

The aim of the study would be to standardize practice in how much epidural catheter is threaded into the epidural space.

ELIGIBILITY:
Inclusion Criteria:

* All women aged 18 years and above.
* In established second stage of labor.
* 3-7 cm dilation at time of insertion.
* Women with BMI < 40 kg/m2

Exclusion Criteria:

* Known contraindication to epidural insertion.
* Inability or unwillingness to provide written consent.
* Previous difficult epidural insertion.
* Previous failed epidural.
* Imminent instrumental or operative delivery.
* Dural puncture.
* Combined spinal epidural analgesia.
* High BMI > 40 kg/m2

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensory block level < T10 | 1 hour
  Sensory block level to ice will be measured 1 hour after the loading dose is administered.
  Yes: inadequate block No: adequate block
Block height discrepancy | 24 hours
  Unilateral block or block height discrepancy of >3 dermatomal levels at any time prior to delivery.
  Yes: inadequate block No: adequate block
Re-siting of the epidural | 24 hours
  Re-siting of the epidural at any time during labour will indicate an inadequate block, for any of the following reasons:
  * Inadequate analgesia
  * Persistent unilateral block
  * Persistent intravascular placement
  * Extensive motor block
  * Hypotension
  * High block
Adjustment of catheter length | 24 hours
  Adjustment of catheter length at any time during labour would also indicate an inadequate block.
Abandonment of epidural or substitute for alternative method of analgesia after initial failure: questionnaire | 24 hours
  The epidural analgesia will also be considered inadequate if the procedure is abandoned or another method of analgesia is used. This will be recorded by the anesthesiologist.

SECONDARY OUTCOMES:
Pain score >3 at any time during labour: questionnaire | 24 hours
  A verbal numerical rating score (VNRS) greater than 3, where 0=no pain and 10=worst pain ever.
Number of epidural top-ups administered by the nursing team | 24 hours
  The number of times the labour and delivery nurse has to administer a top-up of the epidural.
Number of epidural top-ups administered by the anesthesiologist | 24 hours
  The number of times the anesthesiologist has to administer a top-up of the epidural.
Pain scores recorded throughout labour: questionnaire | 24 hours
  A verbal numerical rating score (VNRS), where 0=no pain and 10=worst pain ever. A verbal numerical rating score (VNRS) greater than 3, where 0=no pain and 10=worst pain ever.
Hourly sensory block height assessment | 24 hours
  Hourly sensory block height assessment, using sensation to ice. This is recorded hourly as standard practice.
Incidence of intravascular epidural placement | 24 hours
  Any incidence of intravascular epidural placement during labour will be recorded.
Incidence of catheter dislodgement | 24 hours
  Any incidence of catheter dislodgement during labour will be recorded.
Motor block using Bromage scale | 24 hours
  Bromage scale will be recorded hourly as standard practice.
  * 3: Unable to move feet or knees
  * 2: Able to move feet only
  * 1: Able to just move knees
  * 0: Full flexion of knees and feet
Presence of paresthesia on insertion. | 1 hour
  Any presence of paresthesia on insertion will be recorded.
Adequacy of conversion to surgical block if required for cesarean delivery: questionnaire | 24 hours
  Adequacy of conversion to surgical block in cases requiring cesarean deliveries for failed labor or fetal issues. This will be recorded by the anesthesiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No